CLINICAL TRIAL: NCT01228227
Title: High Loading ROsuvastatin Pretreatment in Patients Undergoing Elective PCI to Reduce the Incidence of MyocArdial Periprocedural Necrosis : Comparison With Atorvastatin High Dose Reloading.
Brief Title: ROsuvastatin Pretreatment to Reduce MyocArdial Periprocedural Necrosis:Comparison With Atorvastatin Reloading
Acronym: ROMAIIReload
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gennaro Sardella (Other)
Responsible Party: Sponsor-Investigator, Gennaro Sardella, Associate Professor in Cardiology, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROMA II
Record Dates: First submitted 2010-10-18; First posted 2010-10-26 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Assess the Periprocedural Myocardial Necrosis
Keywords: Myonecrosis; Percutaneous Angioplasty; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ROSUVASTATIN (Active Comparator)
  Interventions: Drug: ROSUVASTATIN 40 mg
- ATORVASTATIN (Experimental)
  Interventions: Drug: ATORVASTATIN 80 mg

INTERVENTIONS:
Drug: ATORVASTATIN 80 mg — reload of Atorvastatin 80 mg before the procedure
  Arms: ATORVASTATIN
Drug: ROSUVASTATIN 40 mg — reload of rosuvastatin 40 mg before the procedure
  Arms: ROSUVASTATIN

SUMMARY:
An increase in cardiac biomarkers has been shown to occur in 5% to 30% of patients after otherwise successful percutaneous coronary interventions (PCIs)(1) Apart from side-branch occlusion, intimal dissection and coronary spasm, a possible aetiology of myonecrosis after PCI might be distal embolization of atherogenic materials from plaque disruption,(2 )causing obstruction of blood flow at capillary level resulting in micro-infarction.(3,4 )Recent studies have suggested that pretreatment with Atorvastatin may be associated with a reduction in infarct size after elective PCI. (5-7 ). Actually the standard pretreatment in patients undergoing elective coronary-PCI and already treated with aspirin is clopidogrel loading dose administration before procedure.(8,9)The investigators compared a high (80mg) re-loading dose of Atorvastatin with a high loading dose of Rosuvastatin (40 mg) both administered within 24h before the procedure in reducing the rate of periprocedural MI. Therefore, the investigators will conduct a single center, prospective randomized study to assess whether a single, high (80mg) loading (within 24h)dose of Atorvastatin compared with a single loading dose of Rosuvastatin (20 mg) is effective in preventing elevation of biomarkers of MI after elective coronary stent implantation. We evaluate the incidence of MACCE(occurring of cardiac death, myocardial infarction (including periprocedural myonecrosis) and stroke at 30 days 6 and 12 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients with stable angina

Exclusion Criteria:

Baseline myocardial enzyme rise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Myocardial enzymes arise | 12- 24 hours

SECONDARY OUTCOMES:
MACCE | 1-6-12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I, Roma, Roma, Italy